CLINICAL TRIAL: NCT04950686
Title: The Community College Health Study: A Study of Long-term Efficacy and Mechanisms Underlying the Impact of a Web-based Sexual and Relationship Health Promotion Program With Young Adult Community College Students
Brief Title: Study of Long-term Efficacy and Mechanisms Underlying the Impact of a Web-based Sexual and Relationship Health Promotion Program With Young Adult Community College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovation Research & Training (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CCHealthStudy-R01-20-007; R01HD099134 (NIH)
Record Dates: First submitted 2021-05-03; First posted 2021-07-06 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Sexual Behavior; Sexual Assault; Violence, Domestic
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be informed which conditions are considered intervention versus control. All measures are assessed using a web-based data collection system rather than a human outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention - Media Aware for Young Adults (Experimental): This arm will receive Media Aware for Young Adults between the pretest and posttest questionnaire. Media Aware for Young Adults is a web-based sexual and relationship health promotion program that uses a media literacy education (MLE) approach. The program is self-paced and includes four modules.
  Interventions: Behavioral: Media Aware for Young Adults
- Active Control - Health Aware for Young Adults (Active Comparator): This arm will receive Health Aware for Young Adults in between the pretest and posttest questionnaire. Health Aware for Young Adults is a web-based sexual and relationship health promotion program. The program contains the same health content as Media Aware for Young Adults but without the media literacy education components. The program is self-paced and includes four modules.
  Interventions: Behavioral: Health Aware for Young Adults
- Delayed Intervention Control (No Intervention): Participants in this condition will not receive a sexual or relationship health promotion program until after the 12-month follow-up survey. After that survey is complete, they will receive access to the Media Aware for Young Adults program.

INTERVENTIONS:
Behavioral: Media Aware for Young Adults — Media Aware for Young Adults is a web-based sexual and relationship health promotion program designed for young adults that uses a media literacy education (MLE) approach.
  Arms: Intervention - Media Aware for Young Adults
Behavioral: Health Aware for Young Adults — Media Aware for Young Adults is a web-based sexual and relationship health promotion program designed for young adults.
  Arms: Active Control - Health Aware for Young Adults

SUMMARY:
Community college students are an underserved and at-risk population in terms of their sexual and relationship health. This is a three-arm randomized control trial to evaluate the long-term efficacy of a web-based sexual and relationship health promotion program among U.S. community college students (expected N = 2010) and explore the mechanisms underlying the program efficacy.

DETAILED DESCRIPTION:
Community college students are an underserved and at-risk population in terms of their sexual and relationship health. One promising avenue for improving sexual decision making among this population is media literacy education (MLE). Though studies show MLE is an effective approach to sexual health promotion there is a need to better understand the mechanisms by which MLE programs impact health outcomes. The ultimate goals of this study are to 1) advance theoretical frameworks of media literacy to better understand the underlying mechanisms that lead to sexual health behavior change and 2) enhance the sexual and relationship health of community college students by identifying successful methods of health promotion and strategies to implement health programs at community colleges. This study is a three-arm randomized control trial (RCT) with 2010 community college students (ages 18-19) from 30 colleges across the U.S. All components of this study (i.e., interventions, surveys) are web-based.

Participating students will be randomized to one of three conditions: 1) students who receive a sexual health program grounded in MLE (Media Aware); 2) students who receive a sexual health program with no MLE; and 3) a wait-list control group. Participants will complete pretest, posttest, 6-month follow-up, and 12-month follow-up surveys to examine changes across the three groups in our primary outcomes (e.g., risky sexual behavior) and secondary outcomes (e.g., sexual health knowledge, rape myth acceptance, perceived realism of media messages).

ELIGIBILITY:
Inclusion Criteria:

* Students must be 18 or 19 years of age.
* Students must attend one of the community colleges from which this study is recruiting participants.
* Students must have an email address to receive study communication.
* Students must have access to a computer, tablet, or phone device with internet access as the questionnaires and programs are web-based.
* Students must be able to speak and read English because the study materials (e.g., questionnaires, programs) are in English.

Exclusion Criteria:

-

Ages: 18 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2184 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2024-03-24 (Actual); Study Completion 2024-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy M Scull, PhD, Principal Investigator — innovation Research and Training
Locations (1):
- innovation Research and Training, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2184 students consented to participate in the study and were sent the pretest.1647 students completed pretest. Students who did not complete pretest, were dropped from the study and were not considered part of the study sample.
Period: Overall Study
Arm/Group | Intervention - Media Aware for Young Adults | Active Control - Health Aware for Young Adults | Delayed Intervention Control
Started (Started = Completed pretest) | 551 | 508 | 588
Completed Posttest | 376 | 348 | 461
Completed 6-month Follow-up | 342 | 335 | 402
Completed 12-month Follow-up | 330 | 317 | 390
Completed (Per the study protocol, participants did not have to complete every timepoint to remain enrolled in the study. Therefore, the "completed" number listed is the number of participants in each condition that completed the 12-month follow-up (final timepoint).) | 330 | 317 | 390
Not Completed | 221 | 191 | 198

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention - Media Aware for Young Adults | Active Control - Health Aware for Young Adults | Delayed Intervention Control | Total
Number analyzed (Participants) | 551 | 508 | 588 | 1647
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 551 | 508 | 588 | 1647
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.50 (0.5) | 18.51 (0.5) | 18.45 (0.5) | 18.49 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Not all participants reported male or female as their sex.
  Participants
    number analyzed (Participants) | 512 | 490 | 544 | 1546
    Female | 341 | 318 | 338 | 997
    Male | 171 | 172 | 206 | 549
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 132 | 181 | 213 | 526
  Not Hispanic or Latino | 419 | 327 | 375 | 1121
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 8 | 19 | 35
  Asian | 110 | 27 | 44 | 181
  Native Hawaiian or Other Pacific Islander | 5 | 5 | 6 | 16
  Black or African American | 77 | 56 | 66 | 199
  White | 242 | 335 | 323 | 900
  More than one race | 63 | 32 | 63 | 158
  Unknown or Not Reported | 46 | 45 | 67 | 158
Region of Enrollment [Number; unit: participants]
  United States | 551 | 508 | 588 | 1647

OUTCOME MEASURES:

1. Primary Outcome: Relationship Satisfaction
Description: Relationship satisfaction will be assessed using 7-items (e.g., "How well does your partner meet your needs?") rated on a 5-point Likert-type scale from 1 (poorly) to 5 (extremely well); higher scores indicate greater relationship satisfaction; range = 1-5; higher scores indicate a more favorable outcome. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Population: Question only asked of participants in a relationship.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Active Comparator: Active Control - Health Aware for Young Adults: This arm will receive Health Aware for Young Adults in between the pretest and posttest questionnaire. Health Aware for Young Adults is a web-based sexual and relationship health promotion program. The program contains the same health content as Media Aware for Young Adults but without the media literacy education components. The program is self-paced and includes four modules.
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 214 | 251 | 214
score on a scale | 4.22 (0.06) | 4.21 (0.05) | 4.29 (0.06)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — To examine intervention effects on primary outcomes, we used multilevel regression in intent-to-treat analyses. Posttest scores were regressed onto pretest scores, covariates, and the treatment effect. School identifier (ID) was included as a random intercept to adjust for data nesting; p = 0.983, Mixed Models Analysis; Mean Difference (Net) = 0.002, Standard Error of Mean .08
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.465, Mixed Models Analysis; Mean Difference (Net) = -0.06, Standard Error of Mean 0.09

2. Primary Outcome: Relationship Satisfaction
Description: as for outcome 1
Time Frame: 6-month follow-up
Population: Question only asked of participants in a relationship.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 201 | 233 | 194
score on a scale | 4.17 (.07) | 4.23 (.06) | 4.25 (0.08)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — To examine intervention effects on primary outcomes, we used multilevel regression in intent-to-treat analyses. Posttest scores were regressed onto pretest scores, covariates, and the treatment effect. School ID was included as a random intercept to adjust for data nesting; p = 0.579, Mixed Models Analysis; Mean Difference (Net) = -0.05, Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.536, Mixed Models Analysis; Median Difference (Net) = -0.07, Standard Error of Mean 0.12

3. Primary Outcome: Relationship Satisfaction
Description: as for outcome 1
Time Frame: 12-month follow-up
Population: Question only asked of participants in a relationship.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 205 | 225 | 201
score on a scale | 4.22 (0.09) | 4.25 (0.07) | 4.22 (0.10)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.745, Mixed Models Analysis; Mean Difference (Net) = -0.04, Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.972, Mixed Models Analysis; Mean Difference (Net) = 0.005, Standard Error of Mean 0.14

4. Primary Outcome: Percentage of Participants With Relationship Violence Perpetration
Description: 10-items (e.g., "I spoke to my partner in a hostile or mean tone of voice."); Participants were asked to rate how often these things happened with their current or ex-dating partner on a 4-point Likert-type scale from 1 (never) to 4 (often); higher scores indicate more frequent relationship violence; range = 1-4. [Given lack of variability, this measure was dichotomized so 0 equals no violence and 1 equals any violence.]
Time Frame: posttest (4-weeks after pretest)
Population: Only asked of participants in a relationship. This analysis was conducted using multiple imputed data. Therefore, the percentage values will not yield a whole participant because results are pooled between multiple imputations.
Measure: Number; unit: percentage of participants
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 214 | 251 | 214
percentage of participants | 39 | 38 | 38
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.682, Mixed Models Analysis; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.24 to 5.25]
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.630, Mixed Models Analysis; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.28 to 4.69]

5. Primary Outcome: Percentage of Participants With Relationship Violence Perpetration
Description: as for outcome 4
Time Frame: 6-month follow-up
Population: Asked of participants in a relationship. This analysis was conducted using multiple imputed data. Therefore, the percentage values will not yield a whole participant because results are pooled between multiple imputations.
Measure: Number; unit: percentage of participants
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 201 | 233 | 194
percentage of participants | 43 | 40 | 37
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.418, Mixed Models Analysis; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.12 to 12.82]
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.194, Mixed Models Analysis; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.13 to 17.29]

6. Primary Outcome: Percentage of Participants With Relationship Violence Perpetration
Description: as for outcome 4
Time Frame: 12-month follow-up
Population: Asked of participants in a relationship.
Measure: Number; unit: percentage of participants
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 205 | 225 | 201
percentage of participants | 43 | 45 | 41
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.731, Mixed Models Analysis; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.10 to 8.07]
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.786, Mixed Models Analysis; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.16 to 7.34]

7. Primary Outcome: Percentage of Participants With Relationship Violence Victimization
Description: 10-items (e.g., "My partner spoke to me in a hostile or mean tone of voice"); Participants were asked to rate how often these things happened with their current or ex-dating partner on a 4-point Likert-type scale from 1 (never) to 4 (often); higher scores indicate more frequent relationship violence; range = 1-4; [Given lack of variability, this measure was dichotomized so 0 equals no violence and 1 equals any violence.]
Time Frame: posttest (4-weeks after pretest)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 214 | 251 | 214
percentage of participants | 38 | 38 | 36
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.710, Mixed Models Analysis; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.16 to 7.49]
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.610, Mixed Models Analysis; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.16 to 8.73]

8. Primary Outcome: Percentage of Participants With Relationship Violence Victimization
Description: as for outcome 7
Time Frame: 6-month follow-up
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 201 | 233 | 194
percentage of participants | 41 | 36 | 39
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.270, Mixed Models Analysis; Odds Ratio (OR) = 1.37, 95% CI 2-sided [.09 to 20.33]
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.465, Mixed Models Analysis; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.08 to 18.57]

9. Primary Outcome: Percentage of Participants With Relationship Violence Victimization
Description: as for outcome 7
Time Frame: 12-month follow-up
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 205 | 225 | 201
percentage of participants | 45 | 46 | 39
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.702, Mixed Models Analysis; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.07 to 11.95]
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.538, Mixed Models Analysis; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.19 to 7.56]

10. Primary Outcome: Risky Sexual Behaviors
Description: 4-items (e.g., How many times have you had oral, vaginal, or anal sex with a casual partner?); Participants were asked to report how many times each behavior happened; higher scores indicate greater sexual risk taking. Responses were open-ended so while the lower limit of the range was assumed to be zero, there was no upper limit imposed on participants.
Time Frame: posttest (4-weeks after pretest)
Population: Only participants who indicated they had had sex responded to these items.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 318 | 375 | 344
score on a scale | 0.36 (0.03) | 0.29 (0.02) | 0.33 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.084, Mixed Models Analysis; Mean Difference (Net) = 0.06, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.501, Mixed Models Analysis; Mean Difference (Net) = 0.03, Standard Error of Mean 0.04

11. Primary Outcome: Risky Sexual Behaviors
Description: as for outcome 10
Time Frame: 6-month follow-up
Population: Only participants who indicated they had had sex responded to these items.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 318 | 375 | 344
score on a scale | 0.41 (0.02) | 0.40 (0.02) | 0.41 (0.02)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.614, Mixed Models Analysis; Mean Difference (Net) = 0.02, Standard Error of Mean 0.03
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.854, Mixed Models Analysis; Mean Difference (Net) = 0.01, Standard Error of Mean 0.03

12. Primary Outcome: Risky Sexual Behaviors
Description: as for outcome 10
Time Frame: 12-month follow-up
Population: Only participants who indicated they had had sex responded to these items.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 318 | 375 | 344
score on a scale | 0.45 (0.02) | 0.42 (0.02) | 0.43 (0.02)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.499, Mixed Models Analysis; Mean Difference (Net) = 0.02, Standard Error of Mean 0.03
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.623, Mixed Models Analysis; Mean Difference (Net) = 0.02, Standard Error of Mean 0.04

13. Primary Outcome: Percentage of Participants That Used Protection at Last Oral Sex
Description: 1-item ("Did you use a condom and/or dental dam the last time you had oral sex?"); participants answered "yes" (1) or "no" (0); Only participants who indicated they had had oral sex responded to this item
Time Frame: posttest (4-weeks after pretest)
Population: Participants who had sex responded to this item. This analysis was conducted using multiple imputed data - the percentage values will not yield a whole participant because results are pooled between multiple imputations.
Measure: Number; unit: percentage of participants
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 269 | 341 | 297
percentage of participants | 19 | 17 | 17
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.618, Mixed Models Analysis; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.14 to 5.15]
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.626, Mixed Models Analysis; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.10 to 14.13]

14. Primary Outcome: Percentage of Participants That Used Protection at Last Oral Sex
Description: as for outcome 13
Time Frame: 6-month follow-up
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 269 | 341 | 297
percentage of participants | 27 | 19 | 26
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = .232, Mixed Models Analysis; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.23 to 9.18]
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.811, Mixed Models Analysis; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.22 to 5.38]

15. Primary Outcome: Percentage of Participants That Used Protection at Last Oral Sex
Description: as for outcome 13
Time Frame: 12-month follow-up
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 269 | 341 | 297
percentage of participants | 26 | 20 | 21
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.427, Mixed Models Analysis; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.16 to 9.94]
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.337, Mixed Models Analysis; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.25 to 7.68]

16. Primary Outcome: Frequency of Use of Protection During Oral Sex
Description: 3-items used to calculate change in frequency of use of protection during oral sex [e.g., "In the past month, how often did you or your partner(s) use a condom or dental dam when having oral sex?"]; items rated on a 4-point Likert-type scale from 1 (never) to 4 (always) and averaged for analyses; higher scores indicate more frequent use of protection; Only participants who indicated they had had oral sex responded to these items.
Time Frame: posttest (4-weeks after pretest)
Population: Only participants who indicated they had had sex responded to these items.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 269 | 341 | 297
score on a scale | 1.73 (0.09) | 1.63 (0.07) | 1.75 (0.08)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.419, Mixed Models Analysis; Mean Difference (Net) = 0.09, Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.808, Mixed Models Analysis; Mean Difference (Net) = 0.03, Standard Error of Mean 0.12

17. Primary Outcome: Frequency of Use of Protection During Oral Sex
Description: as for outcome 16
Time Frame: 6-month follow-up
Population: Only participants who indicated they had had sex responded to these items.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 269 | 341 | 297
score on a scale | 1.82 (0.09) | 1.76 (0.07) | 1.79 (0.08)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.616, Mixed Models Analysis; Mean Difference (Net) = 0.06, Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.486, Mixed Models Analysis; Mean Difference (Net) = 0.08, Standard Error of Mean 0.12

18. Primary Outcome: Frequency of Use of Protection During Oral Sex
Description: as for outcome 16
Time Frame: 12-month follow-up
Population: Only participants who indicated they had had sex responded to these items.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 269 | 341 | 297
score on a scale | 1.71 (0.09) | 1.76 (0.08) | 1.89 (0.09)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.638, Mixed Models Analysis; Mean Difference (Net) = -0.06, Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.226, Mixed Models Analysis; Mean Difference (Net) = -0.17, Standard Error of Mean 0.14

19. Primary Outcome: Frequency of Condom Use During Vaginal Sex
Description: 3-items used to calculate change in frequency of condom use during vaginal sex [e.g., "In the past month, how often did you or your partner(s) use a condom when having vaginal sex?"]; items rated on a 4-point Likert-type scale from 1 (never) to 4 (always) and averaged for analyses; higher scores indicate more frequent condom use; Only participants who indicated they had had vaginal sex responded to these items.
Time Frame: posttest (4-weeks after pretest)
Population: Only participants who indicated they had had sex responded to these items.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 248 | 306 | 287
score on a scale | 2.5 (0.11) | 2.43 (0.08) | 2.61 (0.10)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.630, Mixed Models Analysis; Mean Difference (Net) = 0.07, Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.880, Mixed Models Analysis; Mean Difference (Net) = -0.02, Standard Error of Mean 0.15

20. Primary Outcome: Frequency of Condom Use During Vaginal Sex
Description: as for outcome 19
Time Frame: 6-month follow-up
Population: Only participants who indicated they had had sex responded to these items.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 248 | 306 | 287
score on a scale | 2.81 (0.08) | 2.75 (0.07) | 2.83 (0.08)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.569, Mixed Models Analysis; Mean Difference (Net) = 0.06, Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.980, Mixed Models Analysis; Mean Difference (Net) = 0.003, Standard Error of Mean 0.12

21. Primary Outcome: Frequency of Condom Use During Vaginal Sex
Description: as for outcome 19
Time Frame: 12-month follow-up
Population: Only participants who indicated they had had sex responded to these items.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 248 | 306 | 287
score on a scale | 2.70 (0.10) | 2.79 (0.09) | 2.71 (0.08)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.466, Mixed Models Analysis; Mean Difference (Net) = -0.10, Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.990, Mixed Models Analysis; Mean Difference (Net) = -0.002, Standard Error of Mean 0.13

22. Primary Outcome: Frequency of Birth Control Use
Description: 3-items used to calculate change in frequency of birth control use [e.g., "In the past month, how often did you or your partner(s) use one of the following forms of birth control? Birth control pills, The Shot (DepoProvera), The Patch, The Ring (Nuvaring), IUD (Mirena, Paragard, Skyla), The Implant (Implanon, Nexplanon), or other FDA approved methods."]; items rated on a 4-point Likert-type scale from 1 (never) to 4 (always) and averaged for analyses; higher scores indicate more frequent birth control use; Only participants who indicated they had had vaginal sex responded to these items.
Time Frame: posttest (4-weeks after pretest)
Population: Only participants who indicated they had had sex responded to these items.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 248 | 306 | 287
score on a scale | 2.48 (0.10) | 2.47 (0.09) | 2.55 (0.11)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.989, Mixed Models Analysis; Mean Difference (Net) = 0.002, Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.678, Mixed Models Analysis; Mean Difference (Net) = -0.07, Standard Error of Mean 0.16

23. Primary Outcome: Frequency of Birth Control Use
Description: as for outcome 22
Time Frame: 6-month follow-up
Population: Only participants who indicated they had had sex responded to these items.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 248 | 306 | 287
score on a scale | 2.56 (0.11) | 2.81 (0.09) | 2.87 (0.10)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.075, Mixed Models Analysis; Mean Difference (Net) = -0.26, Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.024, Mixed Models Analysis; Mean Difference (Net) = -0.35, Standard Error of Mean 0.15

24. Primary Outcome: Frequency of Birth Control Use
Description: as for outcome 22
Time Frame: 12-month follow-up
Population: Only participants who indicated they had had sex responded to these items.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 248 | 306 | 287
score on a scale | 2.67 (0.12) | 2.83 (0.09) | 2.71 (0.11)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.301, Mixed Models Analysis; Mean Difference (Net) = -0.16, Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.702, Mixed Models Analysis; Mean Difference (Net) = -0.07, Standard Error of Mean 0.17

25. Primary Outcome: Percentage of Participants That Used Contraceptive at Last Vaginal Sex
Description: 1-item ("Did you use any contraceptive method the last time you had vaginal sex?"); participants answered "yes" (1) or "no" (0); Only participants who indicated they had had vaginal sex responded to this item
Time Frame: posttest (4-weeks after pretest)
Population: Participants who had sex responded to this item. Analysis was conducted using multiple imputed data- the percentage values will not yield a whole participant because results are pooled between multiple imputations.
Measure: Number; unit: percentage of participants
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 248 | 306 | 287
percentage of participants | 57 | 62 | 64
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.352, Mixed Models Analysis; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.10 to 6.13]
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.445, Mixed Models Analysis; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.11 to 6.16]

26. Primary Outcome: Percentage of Participants That Used Contraceptives at Last Vaginal Sex
Description: as for outcome 25
Time Frame: 6-month follow-up
Population: as for outcome 25
Measure: Number; unit: percentage of participants
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 248 | 306 | 287
percentage of participants | 51 | 62 | 62
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.039, Mixed Models Analysis; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.12 to 2.60]
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.073, Mixed Models Analysis; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.17 to 2.12]

27. Primary Outcome: Percentage of Participants That Used Contraceptives at Last Vaginal Sex
Description: as for outcome 25
Time Frame: 12-month follow-up
Population: as for outcome 25
Measure: Number; unit: percentage of participants
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 248 | 306 | 287
percentage of participants | 54 | 63 | 62
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.110, Mixed Models Analysis; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.13 to 2.93]
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.174, Mixed Models Analysis; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.11 to 3.78]

28. Primary Outcome: Frequency of Condom Use During Anal Sex
Description: 3-items used to calculate change in frequency of condom use during anal sex [e.g., "In the past month, how often did you or your partner(s) use a condom when having anal sex?"]; items rated on a 4-point Likert-type scale from 1 (never) to 4 (always) and averaged for analyses; higher scores indicate more frequent condom use; Only participants who indicated they had had anal sex responded to these items.
Time Frame: posttest (4-weeks after pretest)
Population: Only participants who indicated they had had anal sex responded to these items.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 75 | 86 | 83
score on a scale | 2.33 (0.24) | 1.94 (0.18) | 2.59 (0.25)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.208, Mixed Models Analysis; Mean Difference (Net) = 0.39, Standard Error of Mean 0.31
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.302, Mixed Models Analysis; Mean Difference (Net) = -0.37, Standard Error of Mean 0.35

29. Primary Outcome: Frequency of Condom Use During Anal Sex
Description: as for outcome 28
Time Frame: 6-month follow-up
Population: Only participants who indicated they had had anal sex responded to these items.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 75 | 86 | 83
score on a scale | 2.59 (0.25) | 2.35 (0.22) | 2.47 (0.19)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.483, Mixed Models Analysis; Mean Difference (Net) = 0.24, Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.933, Mixed Models Analysis; Mean Difference (Net) = 0.03, Standard Error of Mean 0.30

30. Primary Outcome: Frequency of Condom Use During Anal Sex
Description: as for outcome 28
Time Frame: 12-month follow-up
Population: Only participants who indicated they had had anal sex responded to these items.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 75 | 86 | 83
score on a scale | 2.41 (0.24) | 2.46 (0.20) | 2.58 (0.21)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.877, Mixed Models Analysis; Mean Difference (Net) = -0.05, Standard Error of Mean 0.32
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.418, Mixed Models Analysis; Mean Difference (Net) = -0.26, Standard Error of Mean 0.32

31. Primary Outcome: Percentage of Participants That Used a Condom at Last Anal Sex
Description: 1-item ("Did you use a condom during your last anal intercourse?"); participants answered "yes" (1) or "no" (0); Only participants who indicated they had had anal sex responded to this item
Time Frame: posttest (4-weeks after pretest)
Population: Participants who had anal sex responded to this item. Analysis was conducted using multiple imputed data - percentage values will not yield a whole participant because results are pooled between multiple imputations.
Measure: Number; unit: percentage of participants
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 75 | 86 | 83
percentage of participants | 53 | 39 | 44
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.220, Mixed Models Analysis; Odds Ratio (OR) = 2.23, 95% CI 2-sided [0.05 to 98.76]
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.10 to 11.30]

32. Primary Outcome: Percentage of Participants That Used a Condom at Last Anal Sex
Description: as for outcome 31
Time Frame: 6-month follow-up
Population: Participants who had sex responded to this item. Analysis was conducted using multiple imputed data - percentage values will not yield a whole participant because results are pooled between multiple imputations.
Measure: Number; unit: percentage of participants
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 75 | 86 | 83
percentage of participants | 47 | 38 | 39
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.506, Mixed Models Analysis; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.03 to 63.29]
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.04 to 36.32]

33. Primary Outcome: Percentage of Participants That Used a Condom at Last Anal Sex
Description: as for outcome 31
Time Frame: 12-month follow-up
Population: as for outcome 32
Measure: Number; unit: percentage of participants
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 75 | 86 | 83
percentage of participants | 47 | 42 | 43
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.877, Mixed Models Analysis; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.04 to 28.37]
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.02 to 26.92]

34. Secondary Outcome: Perceived Realism of Media Messages
Description: 6-items (e.g., "People my age in the media…have sexual contact as often as average people my age"; rated on a 4-point Likert-type scale from 1 (strongly disagree) to 4 (strongly agree); higher scores indicate participants think media is more realistic, indicating a less favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.18 (0.03) | 2.30 (0.03) | 2.43 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.005, Mixed Models Analysis; Mean Difference (Net) = -0.12, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.00001, Mixed Models Analysis; Mean Difference (Net) = -0.23, Standard Error of Mean 0.05

35. Secondary Outcome: Perceived Realism of Media Messages
Description: as for outcome 34
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.27 (0.04) | 2.32 (0.04) | 2.36 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.314, Mixed Models Analysis; Mean Difference (Net) = -0.05, Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.176, Mixed Models Analysis; Mean Difference (Net) = -0.08, Standard Error of Mean 0.06

36. Secondary Outcome: Perceived Realism of Media Messages
Description: as for outcome 34
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.20 (0.04) | 2.33 (0.03) | 2.38 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.009, Mixed Models Analysis; Mean Difference (Net) = -0.13, Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.008, Mixed Models Analysis; Mean Difference (Net) = -0.17, Standard Error of Mean 0.07

37. Secondary Outcome: Perceived Similarity to Media Messages
Description: 7-items (e.g., "The things I do in my life are similar to what I see in the media"); rated on a 4-point Likert-type scale from 1 (strongly disagree) to 4 (strongly agree); higher scores indicate greater perceived similarity, which is a less favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Active Comparator: Active Control - Health Aware for Young Adults: To examine intervention effects on primary outcomes, we used multilevel regression in intent-to-treat analyses. Posttest scores were regressed onto pretest scores, covariates, and the treatment effect. School identifier (ID) was included as a random intercept to adjust for data nesting.
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.04 (0.03) | 2.09 (0.02) | 2.17 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.132, Mixed Models Analysis; Mean Difference (Net) = -0.05, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.008, Mixed Models Analysis; Mean Difference (Net) = -0.11, Standard Error of Mean 0.04

38. Secondary Outcome: Perceived Similarity to Media Messages
Description: as for outcome 37
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.10 (0.03) | 2.11 (0.03) | 2.15 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.941, Mixed Models Analysis; Mean Difference (Net) = -0.003, Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.569, Mixed Models Analysis; Mean Difference (Net) = -0.03, Standard Error of Mean 0.05

39. Secondary Outcome: Perceived Similarity to Media Messages
Description: as for outcome 37
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.05 (0.03) | 2.09 (0.03) | 2.16 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.354, Mixed Models Analysis; Mean Difference (Net) = -0.04, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.038, Mixed Models Analysis; Mean Difference (Net) = -0.11, Standard Error of Mean 0.05

40. Secondary Outcome: Identification With Media
Description: 3-items (e.g., "I want to do the things that people my age in the media do"); rated on a 4-point Likert-type scale from 1 (strongly disagree) to 4 (strongly agree); higher scores indicate participants identify more with media, which is a less favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.38 (0.04) | 2.41 (0.03) | 2.40 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.501, Mixed Models Analysis; Mean Difference (Net) = -0.03, Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.385, Mixed Models Analysis; Mean Difference (Net) = -0.05, Standard Error of Mean 0.06

41. Secondary Outcome: Identification With Media
Description: as for outcome 40
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.35 (0.05) | 2.45 (0.04) | 2.38 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.095, Mixed Models Analysis; Mean Difference (Net) = -0.11, Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.349, Mixed Models Analysis; Mean Difference (Net) = -0.06, Standard Error of Mean 0.07

42. Secondary Outcome: Identification With Media
Description: as for outcome 40
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.41 (0.05) | 2.42 (0.04) | 2.49 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.846, Mixed Models Analysis; Mean Difference (Net) = -0.01, Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.103, Mixed Models Analysis; Mean Difference (Net) = -0.11, Standard Error of Mean 0.07

43. Secondary Outcome: Media Skepticism
Description: 6-items (e.g., "The media are dishonest about what happens when people drink alcohol"); rated on a 4-point Likert-type scale from 1 (strongly disagree) to 4 (strongly agree); higher scores indicate participants have more media skepticism, which is a more favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.13 (0.04) | 3.12 (0.03) | 3.02 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.864, Mixed Models Analysis; Mean Difference (Net) = 0.01, Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.054, Mixed Models Analysis; Mean Difference (Net) = 0.11, Standard Error of Mean 0.06

44. Secondary Outcome: Media Skepticism
Description: as for outcome 43
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.13 (0.04) | 3.06 (0.03) | 3.00 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.168, Mixed Models Analysis; Mean Difference (Net) = 0.07, Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.063, Mixed Models Analysis; Mean Difference (Net) = 0.11, Standard Error of Mean 0.06

45. Secondary Outcome: Media Skepticism
Description: as for outcome 43
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.06 (0.04) | 3.05 (0.04) | 3.04 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.819, Mixed Models Analysis; Mean Difference (Net) = 0.01, Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.775, Mixed Models Analysis; Mean Difference (Net) = 0.02, Standard Error of Mean 0.06

46. Secondary Outcome: Gender Role Norms
Description: 6-items (e.g., "Raising children is primarily a woman's responsibility"); rated on a 4-point Likert-type scale from 1 (strongly disagree) to 4 (strongly agree); higher scores indicate more traditional gender role norms, which is a less favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 1.52 (0.03) | 1.46 (0.02) | 1.56 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.034, Mixed Models Analysis; Mean Difference (Net) = 0.06, Standard Error of Mean 0.03
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.579, Mixed Models Analysis; Mean Difference (Net) = -0.02, Standard Error of Mean 0.05

47. Secondary Outcome: Gender Role Norms
Description: as for outcome 46
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 1.52 (0.03) | 1.49 (0.03) | 1.54 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.485, Mixed Models Analysis; Mean Difference (Net) = 0.03, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.911, Mixed Models Analysis; Mean Difference (Net) = -0.01, Standard Error of Mean 0.05

48. Secondary Outcome: Gender Role Norms
Description: as for outcome 46
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 1.51 (0.03) | 1.49 (0.03) | 1.55 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.583, Mixed Models Analysis; Mean Difference (Net) = 0.02, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.971, Mixed Models Analysis; Mean Difference (Net) = -0.002, Standard Error of Mean 0.04

49. Secondary Outcome: Rape Myth Acceptance
Description: 13-items (e.g., "If a girl is raped while she is drunk, she is at least somewhat responsible for letting things get out of hand"); rated on a 4-point Likert-type scale from 1 (strongly disagree) to 4 (strongly agree); higher scores indicate greater rape myth acceptance, which is a less favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 1.48 (0.03) | 1.46 (0.02) | 1.52 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.602, Mixed Models Analysis; Mean Difference (Net) = 0.02, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.948, Mixed Models Analysis; Mean Difference (Net) = -0.003, Standard Error of Mean 0.04

50. Secondary Outcome: Rape Myth Acceptance
Description: as for outcome 49
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 1.48 (0.03) | 1.46 (0.03) | 1.49 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.763, Mixed Models Analysis; Mean Difference (Net) = 0.01, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.578, Mixed Models Analysis; Mean Difference (Net) = 0.02, Standard Error of Mean 0.04

51. Secondary Outcome: Rape Myth Acceptance
Description: as for outcome 49
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 1.47 (0.03) | 1.46 (0.03) | 1.48 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.863, Mixed Models Analysis; Mean Difference (Net) = 0.01, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.538, Mixed Models Analysis; Mean Difference (Net) = 0.03, Standard Error of Mean 0.04

52. Secondary Outcome: Efficacy to Intervene as Bystander
Description: 5-items (e.g., "I could talk to a friend who I suspected is in an abusive relationship"); participants rate their confidence that they could do the action on a scale from 0-100; higher scores indicate greater bystander efficacy, which is a more favorable outcome; range = 0-100. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 79.05 (1.07) | 79.67 (0.92) | 79.52 (1.30)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.662, Mixed Models Analysis; Mean Difference (Net) = -0.62, Standard Error of Mean 1.41
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.406, Mixed Models Analysis; Mean Difference (Net) = -1.51, Standard Error of Mean 1.81

53. Secondary Outcome: Efficacy to Intervene as Bystander
Description: as for outcome 52
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 77.23 (1.22) | 79.89 (1.04) | 77.55 (1.25)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.105, Mixed Models Analysis; Mean Difference (Net) = -2.66, Standard Error of Mean 1.64
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.487, Mixed Models Analysis; Mean Difference (Net) = -1.33, Standard Error of Mean 1.91

54. Secondary Outcome: Efficacy to Intervene as Bystander
Description: as for outcome 52
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 76.76 (1.26) | 79.06 (1.13) | 78.01 (1.28)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.171, Mixed Models Analysis; Mean Difference (Net) = -2.30, Standard Error of Mean 1.68
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.278, Mixed Models Analysis; Mean Difference (Net) = -2.06, Standard Error of Mean 1.90

55. Secondary Outcome: Intent to Intervene as Bystander
Description: 4-items (e.g., "Approach a friend if I thought they were in an abusive relationship and let them know that I am here to help"); rated on a 4-point Likert-type scale from 1 (not at all likely) to 4 (extremely likely); higher scores indicate greater intentions to intervene as a bystander, which is a more favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.31 (0.03) | 3.36 (0.03) | 3.30 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.283, Mixed Models Analysis; Mean Difference (Net) = -0.04, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.824, Mixed Models Analysis; Mean Difference (Net) = -0.01, Standard Error of Mean 0.05

56. Secondary Outcome: Intent to Intervene as Bystander
Description: as for outcome 55
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.33 (0.03) | 3.33 (0.03) | 3.30 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.965, Mixed Models Analysis; Mean Difference (Net) = -0.002, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.902, Mixed Models Analysis; Mean Difference (Net) = -0.01, Standard Error of Mean 0.05

57. Secondary Outcome: Intent to Intervene as Bystander
Description: as for outcome 55
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.33 (0.03) | 3.40 (0.03) | 3.29 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.074, Mixed Models Analysis; Mean Difference (Net) = -0.07, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.828, Mixed Models Analysis; Mean Difference (Net) = 0.01, Standard Error of Mean 0.05

58. Secondary Outcome: Sexual Health Knowledge
Description: 23-items (e.g., "True or False: You can tell if someone has an STI by looking at him/her"); For each item, participants who answer correctly will receive a "1" and participants who answer incorrectly will receive a "0"; items will be summed; higher scores indicate greater sexual health knowledge; range = 0-23 The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 17.53 (0.18) | 17.29 (0.16) | 17.42 (0.19)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.336, Mixed Models Analysis; Mean Difference (Net) = 0.24, Standard Error of Mean 0.25
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.902, Mixed Models Analysis; Mean Difference (Net) = 0.03, Standard Error of Mean 0.28

59. Secondary Outcome: Sexual Health Knowledge
Description: 23-items (e.g., "True or False: You can tell if someone has an STI by looking at him/her"); For each item, participants who answer correctly will receive a "1" and participants who answer incorrectly will receive a "0"; items will be summed; higher scores indicate greater sexual health knowledge; range = 0-23. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 17.36 (0.18) | 17.48 (0.15) | 17.61 (0.20)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.629, Mixed Models Analysis; Mean Difference (Net) = -0.12, Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.318, Mixed Models Analysis; Mean Difference (Net) = -0.29, Standard Error of Mean 0.29

60. Secondary Outcome: Sexual Health Knowledge
Description: as for outcome 59
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 17.48 (0.19) | 17.53 (0.16) | 17.74 (0.20)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.863, Mixed Models Analysis; Mean Difference (Net) = -0.04, Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.299, Mixed Models Analysis; Mean Difference (Net) = -0.30, Standard Error of Mean 0.29

61. Secondary Outcome: Attitudes Toward Risky Sexual Behaviors
Description: 5-items (e.g., "It is okay to…have sex with someone who has had many sexual partners"); rated on a 4-point Likert-type scale from 1 (strongly disagree) to 4 (strongly agree); higher scores indicate positive attitudes towards risky sexual behaviors, which is a less favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.22 (0.03) | 2.32 (0.03) | 2.25 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.010, Mixed Models Analysis; Mean Difference (Net) = -0.10, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.119, Mixed Models Analysis; Mean Difference (Net) = -0.07, Standard Error of Mean 0.05

62. Secondary Outcome: Attitudes Toward Risky Sexual Behaviors
Description: as for outcome 61
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.24 (.03) | 2.30 (0.03) | 2.28 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.161, Mixed Models Analysis; Mean Difference (Net) = -0.06, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.087, Mixed Models Analysis; Mean Difference (Net) = -0.09, Standard Error of Mean 0.05

63. Secondary Outcome: Attitudes Toward Risky Sexual Behaviors
Description: as for outcome 61
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.26 (0.04) | 2.25 (0.03) | 2.20 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.810, Mixed Models Analysis; Mean Difference (Net) = 0.01, Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.901, Mixed Models Analysis; Mean Difference (Net) = 0.01, Standard Error of Mean 0.06

64. Secondary Outcome: Attitudes Toward Unprotected Sex
Description: 1-item ["It is okay to…have unprotected sex (not including when people are trying to get pregnant)"]; rated on a 4-point Likert-type scale from 1 (strongly disagree) to 4 (strongly agree); higher scores indicate positive attitudes towards unprotected sex; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 1.96 (0.05) | 2.07 (0.05) | 2.04 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.145, Mixed Models Analysis; Mean Difference (Net) = -0.10, Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.096, Mixed Models Analysis; Mean Difference (Net) = -0.12, Standard Error of Mean 0.07

65. Secondary Outcome: Attitudes Toward Unprotected Sex
Description: as for outcome 64
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 1.98 (0.06) | 2.06 (0.05) | 1.98 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.272, Mixed Models Analysis; Mean Difference (Net) = -0.09, Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.689, Mixed Models Analysis; Mean Difference (Net) = -0.03, Standard Error of Mean 0.08

66. Secondary Outcome: Attitudes Toward Unprotected Sex
Description: as for outcome 64
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.05 (0.06) | 2.06 (0.05) | 2.12 (0.06)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.824, Mixed Models Analysis; Mean Difference (Net) = -0.02, Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.271, Mixed Models Analysis; Mean Difference (Net) = -0.10, Standard Error of Mean 0.09

67. Secondary Outcome: Attitudes Toward Contraception/Protection
Description: 9-items (e.g., "It is wrong to use birth control"); rated on a 4-point Likert-type scale from 1 (strongly disagree) to 4 (strongly agree); higher scores indicate more favorable attitudes towards contraception; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.44 (0.03) | 3.47 (0.02) | 3.42 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.391, Mixed Models Analysis; Mean Difference (Net) = -0.03, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.952, Mixed Models Analysis; Mean Difference (Net) = -0.002, Standard Error of Mean 0.04

68. Secondary Outcome: Attitudes Toward Contraception/Protection
Description: as for outcome 67
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.46 (0.03) | 3.46 (0.03) | 3.37 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.925, Mixed Models Analysis; Mean Difference (Net) = 0.004, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.153, Mixed Models Analysis; Mean Difference (Net) = 0.07, Standard Error of Mean 0.05

69. Secondary Outcome: Attitudes Toward Contraception/Protection
Description: as for outcome 67
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.45 (0.04) | 3.42 (0.03) | 3.37 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.495, Mixed Models Analysis; Mean Difference (Net) = 0.03, Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.229, Mixed Models Analysis; Mean Difference (Net) = 0.07, Standard Error of Mean 0.06

70. Secondary Outcome: Attitudes Toward Communication With Partners and Medical Professionals
Description: 4-items (e.g., "Before deciding to have sex, people should…talk with their partner about HIV/AIDS and other STIs"); rated on a 4-point Likert-type scale from 1 (strongly disagree) to 4 (strongly agree); higher scores indicate positive attitudes towards communication, which is a more favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.45 (0.04) | 3.47 (0.03) | 3.47 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.753, Mixed Models Analysis; Mean Difference (Net) = -0.01, Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.350, Mixed Models Analysis; Mean Difference (Net) = -0.05, Standard Error of Mean 0.05

71. Secondary Outcome: Attitudes Toward Communication With Partners and Medical Professionals
Description: as for outcome 70
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.48 (0.03) | 3.50 (0.03) | 3.46 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.541, Mixed Models Analysis; Mean Difference (Net) = -0.03, Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.887, Mixed Models Analysis; Mean Difference (Net) = -0.01, Standard Error of Mean 0.05

72. Secondary Outcome: Attitudes Toward Communication With Partners and Medical Professionals
Description: as for outcome 70
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.44 (0.03) | 3.48 (0.03) | 3.36 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.375, Mixed Models Analysis; Mean Difference (Net) = -0.04, Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.293, Mixed Models Analysis; Mean Difference (Net) = 0.06, Standard Error of Mean 0.06

73. Secondary Outcome: Descriptive Norms of Unprotected Sex
Description: 1-item (e.g., "What percentage of people your age have had unprotected sex?"); participants write in their estimate of what percentage of their peers are engaging in the behavior; higher scores indicate participants think more of their peers are engaging in unprotected sex; range = 0-100. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 46.97 (1.40) | 52.95 (1.23) | 50.56 (1.54)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.002, Mixed Models Analysis; Mean Difference (Net) = -5.97, Standard Error of Mean 1.89
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.163, Mixed Models Analysis; Mean Difference (Net) = -3.08, Standard Error of Mean 2.21

74. Secondary Outcome: Descriptive Norms of Unprotected Sex
Description: as for outcome 73
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 48.81 (1.46) | 53.90 (1.28) | 52.48 (1.52)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.011, Mixed Models Analysis; Mean Difference (Net) = -5.09, Standard Error of Mean 1.99
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.159, Mixed Models Analysis; Mean Difference (Net) = -3.21, Standard Error of Mean 2.27

75. Secondary Outcome: Descriptive Norms of Unprotected Sex
Description: as for outcome 73
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 50.45 (1.54) | 54.28 (1.32) | 54.40 (1.57)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.064, Mixed Models Analysis; Mean Difference (Net) = -3.83, Standard Error of Mean 2.06
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.137, Mixed Models Analysis; Mean Difference (Net) = -3.37, Standard Error of Mean 2.27

76. Secondary Outcome: Descriptive Norms of Risky Sexual Activity
Description: 5-items (e.g., "What percentage of people your age…have had oral, anal, or vaginal sex with someone who has not been tested for STIs or whose STI status is unknown?"); participants write in their estimate of what percentage of their peers are engaging in each behavior; higher scores indicate participants think more of their peers are engaging in risky contraception use/protection practices; range = 0-100. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 44.21 (1.15) | 49.26 (0.97) | 48.00 (1.23)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.001, Mixed Models Analysis; Mean Difference (Net) = -5.05, Standard Error of Mean 1.52
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.065, Mixed Models Analysis; Mean Difference (Net) = -3.25, Standard Error of Mean 1.76

77. Secondary Outcome: Descriptive Norms of Risky Sexual Activity
Description: as for outcome 76
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 46.70 (1.10) | 50.37 (0.97) | 49.80 (1.27)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.015, Mixed Models Analysis; Mean Difference (Net) = -3.67, Standard Error of Mean 1.51
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.152, Mixed Models Analysis; Mean Difference (Net) = -2.56, Standard Error of Mean 1.78

78. Secondary Outcome: Descriptive Norms of Risky Sexual Activity
Description: as for outcome 76
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 45.33 (1.29) | 49.11 (1.14) | 49.08 (1.31)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.034, Mixed Models Analysis; Mean Difference (Net) = -3.78, Standard Error of Mean 1.78
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.090, Mixed Models Analysis; Mean Difference (Net) = -3.13, Standard Error of Mean 1.84

79. Secondary Outcome: Sex Refusal Self-efficacy
Description: 5-items (e.g., "I can easily say 'no' to someone who is pressuring me to have sex"); rated on a 4-point Likert-type scale from 1 (strongly disagree) to 4 (strongly agree); higher scores indicate greater sex refusal self-efficacy, which is a more favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.19 (0.03) | 3.14 (0.03) | 3.16 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.282, Mixed Models Analysis; Mean Difference (Net) = 0.05, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.532, Mixed Models Analysis; Mean Difference (Net) = 0.03, Standard Error of Mean 0.05

80. Secondary Outcome: Sex Refusal Self-efficacy
Description: as for outcome 79
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.17 (0.04) | 3.20 (0.04) | 3.13 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.675, Mixed Models Analysis; Mean Difference (Net) = -0.02, Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.443, Mixed Models Analysis; Mean Difference (Net) = 0.04, Standard Error of Mean 0.06

81. Secondary Outcome: Sex Refusal Self-efficacy
Description: as for outcome 79
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.18 (0.04) | 3.20 (0.03) | 3.20 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.685, Mixed Models Analysis; Mean Difference (Net) = -0.02, Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.726, Mixed Models Analysis; Mean Difference (Net) = -0.02, Standard Error of Mean 0.06

82. Secondary Outcome: Self-efficacy to Refuse Unprotected Sex
Description: 1-item ("I can easily say 'no' to sex if we do not have protection even if I really want to have sex with that person"); rated on a 4-point Likert-type scale from 1 (strongly disagree) to 4 (strongly agree); higher scores indicate greater self-efficacy to refuse unprotected sex, which is a more favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.19 (0.03) | 3.14 (0.03) | 3.26 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.282, Mixed Models Analysis; Mean Difference (Net) = 0.05, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.591, Mixed Models Analysis; Mean Difference (Net) = -0.03, Standard Error of Mean 0.06

83. Secondary Outcome: Self-efficacy to Refuse Unprotected Sex
Description: as for outcome 82
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.17 (0.04) | 3.20 (0.04) | 3.17 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.675, Mixed Models Analysis; Mean Difference (Net) = -0.02, Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.359, Mixed Models Analysis; Mean Difference (Net) = 0.07, Standard Error of Mean 0.08

84. Secondary Outcome: Self-efficacy to Refuse Unprotected Sex
Description: as for outcome 82
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.18 (0.04) | 3.20 (0.03) | 3.29 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — To examine intervention effects on primary outcomes, we used multilevel regression in intent-to-treat analyses. Posttest scores were regressed onto pretest scores, covariates, and the treatment effect. School ID was included as a random intercept to adjust for data nesting.rt-type scale from 1 (strongly disagree) to 4 (strongly agree); higher scores indicate greater self-efficacy to use a dental dam; range = 1-4; p = 0.685, Mixed Models Analysis; Mean Difference (Net) = -0.02, Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.198, Mixed Models Analysis; Mean Difference (Net) = -0.09, Standard Error of Mean 0.07

85. Secondary Outcome: Self-efficacy to Use a Condom
Description: 1-item (e.g., "I can use a condom correctly or explain to my partner how to use a condom correctly"); rated on a 4-point Likert-type scale from 1 (strongly disagree) to 4 (strongly agree); higher scores indicate greater self-efficacy to use a condom, which is a more favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.28 (0.05) | 3.23 (0.04) | 3.27 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — To examine intervention effects on primary outcomes, we used multilevel regression in intent-to-treat analyses. Posttest scores were regressed onto pretest scores, covariates, and the treatment effect. School ID was included as a random intercept to adjust for data nesting.-type scale from 1 (strongly disagree) to 4 (strongly agree); higher scores indicate greater self-efficacy to use a dental dam; range = 1-4; p = 0.460, Mixed Models Analysis; Mean Difference (Net) = 0.05, Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.822, Mixed Models Analysis; Mean Difference (Net) = 0.01, Standard Error of Mean 0.06

86. Secondary Outcome: Self-efficacy to Use a Condom
Description: as for outcome 85
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.27 (0.05) | 3.25 (0.04) | 3.27 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.671, Mixed Models Analysis; Mean Difference (Net) = 0.03, Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.939, Mixed Models Analysis; Mean Difference (Net) = 0.01, Standard Error of Mean 0.07

87. Secondary Outcome: Self-efficacy to Use a Condom
Description: as for outcome 85
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.29 (0.04) | 3.32 (0.04) | 3.23 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.655, Mixed Models Analysis; Mean Difference (Net) = -0.03, Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.315, Mixed Models Analysis; Mean Difference (Net) = 0.07, Standard Error of Mean 0.07

88. Secondary Outcome: Self-efficacy to Communicate With Partners and Medical Professionals About Sex
Description: 4-items (e.g., "I can discuss preventing STIs with my partner"); rated on a 4-point Likert-type scale from 1 (strongly disagree) to 4 (strongly agree); higher scores indicate greater self-efficacy to communicate, which is a more favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.35 (0.03) | 3.35 (0.03) | 3.35 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.966, Mixed Models Analysis; Mean Difference (Net) = 0.002, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.708, Mixed Models Analysis; Mean Difference (Net) = -0.02, Standard Error of Mean 0.05

89. Secondary Outcome: Self-efficacy to Communicate With Partners and Medical Professionals About Sex
Description: as for outcome 88
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.35 (0.03) | 3.34 (0.03) | 3.32 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.887, Mixed Models Analysis; Mean Difference (Net) = 0.006, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.077, Mixed Models Analysis; Mean Difference (Net) = 0.01, Standard Error of Mean 0.05

90. Secondary Outcome: Self-efficacy to Communicate With Partners and Medical Professionals About Sex
Description: as for outcome 88
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.36 (0.03) | 3.42 (0.03) | 3.34 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.217, Mixed Models Analysis; Mean Difference (Net) = -0.05, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.879, Mixed Models Analysis; Mean Difference (Net) = 0.01, Standard Error of Mean 0.05

91. Secondary Outcome: Risky Sexual Behavior Intentions
Description: 5-items (e.g., "In the next 6 months, how likely is it that you will have oral, anal, or vaginal sex with a casual partner"); rated on a 4-point Likert-type scale from 1 (not at all likely) to 4 (extremely likely); higher scores indicate greater intentions to engage in risky sexual behaviors, which is a less favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 1.79 (0.03) | 1.80 (0.03) | 1.79 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.866, Mixed Models Analysis; Mean Difference (Net) = -0.01, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.695, Mixed Models Analysis; Mean Difference (Net) = 0.02, Standard Error of Mean 0.06

92. Secondary Outcome: Risky Sexual Behavior Intentions
Description: as for outcome 91
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 1.79 (0.04) | 1.80 (0.04) | 1.86 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.940, Mixed Models Analysis; Mean Difference (Net) = -0.004, Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.451, Mixed Models Analysis; Mean Difference (Net) = -0.05, Standard Error of Mean 0.06

93. Secondary Outcome: Risky Sexual Behavior Intentions
Description: as for outcome 91
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 1.78 (0.04) | 1.82 (0.04) | 1.90 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.442, Mixed Models Analysis; Mean Difference (Net) = -0.04, Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.082, Mixed Models Analysis; Mean Difference (Net) = -0.11, Standard Error of Mean 0.06

94. Secondary Outcome: Intentions to Have Unprotected Sex
Description: 1-item ("In the next 6 months, how likely is it that you will…have unprotected sex?"); rated on a 4-point Likert-type scale from 1 (not at all likely) to 4 (extremely likely); higher scores indicate greater intentions to have unprotected sex, which is a less favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 1.88 (0.05) | 1.96 (0.04) | 1.91 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.236, Mixed Models Analysis; Mean Difference (Net) = -0.07, Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.674, Mixed Models Analysis; Mean Difference (Net) = -0.03, Standard Error of Mean 0.08

95. Secondary Outcome: Intentions to Have Unprotected Sex
Description: as for outcome 94
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 1.92 (0.05) | 2.03 (0.05) | 1.96 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.135, Mixed Models Analysis; Mean Difference (Net) = -0.11, Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.500, Mixed Models Analysis; Mean Difference (Net) = -0.05, Standard Error of Mean 0.08

96. Secondary Outcome: Intentions to Have Unprotected Sex
Description: as for outcome 94
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 1.98 (0.06) | 1.98 (0.06) | 2.08 (0.06)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.956, Mixed Models Analysis; Mean Difference (Net) = 0.005, Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.214, Mixed Models Analysis; Mean Difference (Net) = -0.11, Standard Error of Mean 0.09

97. Secondary Outcome: Intentions to Use a Condom
Description: 1-item (e.g., "If you were to decide to have sexual intercourse in the next 6 months, how likely would you be to use a condom?"); rated on a 4-point Likert-type scale from 1 (not at all likely) to 4 (extremely likely); higher scores indicate greater intentions to use protection/contraception, which is a more favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.22 (0.05) | 3.16 (0.04) | 3.22 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.337, Mixed Models Analysis; Mean Difference (Net) = 0.06, Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.957, Mixed Models Analysis; Mean Difference (Net) = 0.004, Standard Error of Mean 0.07

98. Secondary Outcome: Intentions to Use a Condom
Description: as for outcome 97
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.25 (0.06) | 3.10 (0.05) | 3.21 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.086, Mixed Models Analysis; Mean Difference (Net) = 0.14, Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.515, Mixed Models Analysis; Mean Difference (Net) = 0.05, Standard Error of Mean 0.08

99. Secondary Outcome: Intentions to Use a Condom
Description: as for outcome 97
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.10 (0.06) | 3.15 (0.05) | 3.07 (0.06)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.597, Mixed Models Analysis; Mean Difference (Net) = -0.04, Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.551, Mixed Models Analysis; Mean Difference (Net) = 0.05, Standard Error of Mean 0.09

100. Secondary Outcome: Intentions to Communicate With Partners and Medical Professionals About Sex
Description: 6-items (e.g., "If you were to decide to engage in sexual activity with a new partner in the next 6 months, how likely would you be to…talk with a partner about HIV/AIDS or other STIs?"); rated on a 4-point Likert-type scale from 1 (not at all likely) to 4 (extremely likely); higher scores indicate greater intentions to communicate, which is a more favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.07 (0.03) | 3.09 (0.03) | 3.13 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.634, Mixed Models Analysis; Mean Difference (Net) = -0.02, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.308, Mixed Models Analysis; Mean Difference (Net) = -0.05, Standard Error of Mean 0.05

101. Secondary Outcome: Intentions to Communicate With Partners and Medical Professionals About Sex
Description: as for outcome 100
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.11 (0.04) | 3.06 (0.04) | 3.09 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.415, Mixed Models Analysis; Mean Difference (Net) = 0.05, Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.721, Mixed Models Analysis; Mean Difference (Net) = 0.02, Standard Error of Mean 0.06

102. Secondary Outcome: Intentions to Communicate With Partners and Medical Professionals About Sex
Description: as for outcome 100
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.05 (0.05) | 3.13 (0.04) | 3.12 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.261, Mixed Models Analysis; Mean Difference (Net) = -0.07, Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.369, Mixed Models Analysis; Mean Difference (Net) = -0.06, Standard Error of Mean 0.06

103. Secondary Outcome: Willingness to Have Unprotected Sex
Description: 1-item (e.g., "Suppose you were with your boyfriend/girlfriend/partner. He/she wants to have sex, but neither of you have any form of protection. In this situation, how willing would you be to go ahead and have sex anyway?";); rated on a 4-point Likert-type scale from 1 (very unwilling) to 4 (very willing); higher scores indicate greater willingness to have unprotected sex, which is a less favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.28 (0.04) | 2.37 (0.04) | 2.24 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.124, Mixed Models Analysis; Mean Difference (Net) = -0.09, Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.794, Mixed Models Analysis; Mean Difference (Net) = 0.02, Standard Error of Mean 0.06

104. Secondary Outcome: Willingness to Have Unprotected Sex
Description: as for outcome 103
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.24 (0.05) | 2.41 (0.04) | 2.34 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.011, Mixed Models Analysis; Mean Difference (Net) = -0.17, Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.068, Mixed Models Analysis; Mean Difference (Net) = -0.13, Standard Error of Mean 0.07

105. Secondary Outcome: Willingness to Have Unprotected Sex
Description: as for outcome 103
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.34 (0.06) | 2.38 (0.05) | 2.38 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.585, Mixed Models Analysis; Mean Difference (Net) = -0.04, Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.338, Mixed Models Analysis; Mean Difference (Net) = -0.07, Standard Error of Mean 0.08

106. Secondary Outcome: Willingness to Engage in Risky Sexual Behaviors
Description: 5-items (e.g., "Suppose you wanted to have sex with someone but you did not know their STI status. In this situation, how willing would you be to have sex anyway?"); rated on a 4-point Likert-type scale from 1 (very unwilling) to 4 (very willing); higher scores indicate greater willingness to engage in risky sexual behaviors, which is a less favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 1.90 (0.03) | 1.94 (0.03) | 1.88 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.259, Mixed Models Analysis; Mean Difference (Net) = -0.05, Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.950, Mixed Models Analysis; Mean Difference (Net) = -0.003, Standard Error of Mean 0.05

107. Secondary Outcome: Willingness to Engage in Risky Sexual Behaviors
Description: as for outcome 106
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 1.91 (0.04) | 1.95 (0.03) | 1.92 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.411, Mixed Models Analysis; Mean Difference (Net) = -0.04, Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.491, Mixed Models Analysis; Mean Difference (Net) = -0.03, Standard Error of Mean 0.05

108. Secondary Outcome: Willingness to Engage in Risky Sexual Behaviors
Description: as for outcome 106
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 1.93 (0.03) | 1.90 (0.03) | 1.89 (0.03)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.498, Mixed Models Analysis; Mean Difference (Net) = 0.03, Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.573, Mixed Models Analysis; Mean Difference (Net) = 0.03, Standard Error of Mean 0.05

109. Secondary Outcome: Advertisement Deconstruction Skills
Description: Participants are shown an advertisement and asked to describe it in detail including noting marketing strategies and any missing information (e.g., How are advertisers trying to get someone to buy this product?). Qualitative responses to the questions are coded by trained project staff members once inter-coder reliability is established, and scores represent the extent to which participants identify the implied message of the advertisement. Range: 0-3. Higher scores indicate a more favorable outcome. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Population: Only includes participants who provided data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 369 | 460 | 354
score on a scale | 1.45 (0.05) | 1.36 (0.05) | 1.20 (0.07)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.128, Mixed Models Analysis; Mean Difference (Net) = 0.09, Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.013, Mixed Models Analysis; Mean Difference (Net) = 0.21, Standard Error of Mean 0.08

110. Secondary Outcome: Injunctive Norms - Most People
Description: 3-items (e.g., "Most people believe that it is okay for people my age to have unprotected sex"); rated on a 4-point Likert-type scale from 1 (strongly disagree) to 4 (strongly agree); higher scores indicate riskier injunctive norms, which is a less favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.16 (0.05) | 2.16 (0.04) | 2.15 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.999, Mixed Models Analysis; Mean Difference (Net) = -0.0001, Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — This arm will receive Health Aware for Young Adults in between the pretest and posttest questionnaire. Health Aware for Young Adults is a web-based sexual and relationship health promotion program. The program contains the same health content as Media Aware for Young Adults but without the media literacy education components. The program is self-paced and includes four modules; p = 0.638, Mixed Models Analysis; Mean Difference (Net) = 0.04, Standard Error of Mean 0.08

111. Secondary Outcome: Injunctive Norms - Most People
Description: as for outcome 110
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.26 (0.05) | 2.25 (0.04) | 2.20 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.841, Mixed Models Analysis; Mean Difference (Net) = 0.01, Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.270, Mixed Models Analysis; Mean Difference (Net) = 0.08, Standard Error of Mean 0.08

112. Secondary Outcome: Injunctive Norms - Most People
Description: as for outcome 110
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.25 (0.06) | 2.24 (0.05) | 2.27 (0.06)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.940, Mixed Models Analysis; Mean Difference (Net) = 0.01, Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.992, Mixed Models Analysis; Mean Difference (Net) = -0.001, Standard Error of Mean 0.09

113. Secondary Outcome: Injunctive Norms - Friends
Description: 1 item ("My friends think I should use protection when I have sex"); rated on a 4-point Likert-type scale from 1 (strongly disagree) to 4 (strongly agree); higher scores less risky injunctive norms, which is a more favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.27 (0.04) | 3.31 (0.04) | 3.35 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.470, Mixed Models Analysis; Mean Difference (Net) = -0.04, Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.130, Mixed Models Analysis; Mean Difference (Net) = -0.09, Standard Error of Mean 0.06

114. Secondary Outcome: Injunctive Norms - Friends
Description: as for outcome 113
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.30 (0.06) | 3.30 (0.05) | 3.32 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.931, Mixed Models Analysis; Mean Difference (Net) = -0.01, Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.666, Mixed Models Analysis; Mean Difference (Net) = -0.03, Standard Error of Mean 0.07

115. Secondary Outcome: Injunctive Norms - Friends
Description: as for outcome 113
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.29 (0.05) | 3.30 (0.04) | 3.30 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.822, Mixed Models Analysis; Mean Difference (Net) = -0.02, Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.721, Mixed Models Analysis; Mean Difference (Net) = -0.03, Standard Error of Mean 0.07

116. Secondary Outcome: Descriptive Norms - People Like me
Description: 1-item ("Most people like me use protection when they have sex"); rated on a 4-point Likert-type scale from 1 (strongly disagree) to 4 (strongly agree); higher scores less risky descriptive norms, which is a more favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.15 (0.04) | 3.12 (0.04) | 3.14 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.540, Mixed Models Analysis; Mean Difference (Net) = 0.03, Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.956, Mixed Models Analysis; Mean Difference (Net) = 0.003, Standard Error of Mean 0.06

117. Secondary Outcome: Descriptive Norms - People Like me
Description: as for outcome 116
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.21 (0.05) | 3.13 (0.04) | 3.11 (0.04)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.175, Mixed Models Analysis; Mean Difference (Net) = 0.09, Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.136, Mixed Models Analysis; Mean Difference (Net) = 0.09, Standard Error of Mean 0.06

118. Secondary Outcome: Descriptive Norms - People Like me
Description: as for outcome 116
Time Frame: 12-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 3.16 (0.05) | 3.15 (0.04) | 3.14 (0.05)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.829, Mixed Models Analysis; Mean Difference (Net) = 0.01, Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.748, Mixed Models Analysis; Mean Difference (Net) = 0.02, Standard Error of Mean 0.07

119. Secondary Outcome: Frequency of Communication With Sexual Partner
Description: 1 item used to calculate change in frequency of sexual communication with a partner(s) [e.g., "In the past month, how often did you talk to your partner(s) about using condoms and/or other forms of contraception before engaging in sexual activity?"]; items rated on a 4-point Likert-type scale from 1 (never) to 4 (always); higher scores indicate more frequent communication, which is a more favorable outcome. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Population: Question only asked of participants who were sexually active.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 318 | 375 | 344
score on a scale | 2.72 (0.09) | 2.81 (0.08) | 2.81 (0.09)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.490, Mixed Models Analysis; Mean Difference (Net) = -0.08, Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.831, Mixed Models Analysis; Mean Difference (Net) = -0.03, Standard Error of Mean 0.13

120. Secondary Outcome: Frequency of Communication With Sexual Partner
Description: as for outcome 119
Time Frame: 6-month follow-up
Population: Question only asked of participants who were sexually active.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 318 | 375 | 344
score on a scale | 3.22 (0.07) | 3.13 (0.06) | 3.14 (0.07)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.350, Mixed Models Analysis; Mean Difference (Net) = 0.09, Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.235, Mixed Models Analysis; Mean Difference (Net) = 0.12, Standard Error of Mean 0.10

121. Secondary Outcome: Frequency of Communication With Sexual Partner
Description: as for outcome 119
Time Frame: 12-month follow-up
Population: Question only asked of participants who were sexually active.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 318 | 375 | 344
score on a scale | 3.21 (0.08) | 3.17 (0.07) | 3.11 (0.08)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.682, Mixed Models Analysis; Mean Difference (Net) = 0.04, Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.373, Mixed Models Analysis; Mean Difference (Net) = 0.10, Standard Error of Mean 0.11

122. Secondary Outcome: Percentage of Participants That Communicated With a Doctor
Description: 1-item used to calculate change in whether participants communicated with a doctor about sex ["In the past month, had you talked to a doctor or other medical professional about sex, contraception, and/or relationships?"]; participants answered "yes" (1) or "no" (0)
Time Frame: posttest (4-weeks after pretest)
Population: Analysis was conducted using multiple imputed data - percentage values will not yield a whole participant because results are pooled between multiple imputations.
Measure: Number; unit: percentage of participants
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
percentage of participants | 23 | 20 | 28
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.242, Mixed Models Analysis; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.24 to 6.63]
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.207, Mixed Models Analysis; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.11 to 5.72]

123. Secondary Outcome: Percentage of Participants That Communicated With a Doctor
Description: as for outcome 122
Time Frame: 6-month follow-up
Population: as for outcome 122
Measure: Number; unit: percentage of participants
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
percentage of participants | 51 | 55 | 53
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.576, Mixed Models Analysis; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.51 to 1.52]
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.888, Mixed Models Analysis; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.46 to 2.03]

124. Secondary Outcome: Percentage of Participants That Communicated With a Doctor
Description: 1 item used to calculate change in whether participants communicated with a doctor about sex ["In the past month, had you talked to a doctor or other medical professional about sex, contraception, and/or relationships?"]; participants answered "yes" (1) or "no" (0)
Time Frame: 12-month follow-up
Population: This analysis was conducted using multiple imputed data. Therefore, the percentage values will not yield a whole participant because results are pooled between multiple imputations.
Measure: Number; unit: percentage of participants
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
percentage of participants | 54 | 57 | 54
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.467, Mixed Models Analysis; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.22 to 3.45]
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.888, Mixed Models Analysis; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.46 to 2.03]

125. Secondary Outcome: Self-efficacy to Use a Dental Dam
Description: 1-item (e.g., "I can use a dental dam correctly or explain to my partner how to use a dental dam correctly"); rated on a 4-point Likert-type scale from 1 (strongly disagree) to 4 (strongly agree); higher scores indicate greater self-efficacy to use a dental dam, which is a more favorable outcome; range = 1-4. The overall number of participants analyzed in each Arm/Group includes all participants who completed pretest. Posttest data was imputed for participants that were present at pretest but not at posttest.
Time Frame: posttest (4-weeks after pretest)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.46 (0.05) | 2.22 (0.04) | 2.40 (0.07)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.0003, Mixed Models Analysis; Mean Difference (Net) = 0.24, Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.432, Mixed Models Analysis; Mean Difference (Net) = 0.07, Standard Error of Mean 0.09

126. Secondary Outcome: Self-efficacy to Use a Dental Dam
Description: as for outcome 125
Time Frame: 6 month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.43 (0.06) | 2.26 (0.05) | 2.40 (0.06)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.031, Mixed Models Analysis; Mean Difference (Net) = 0.16, Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.794, Mixed Models Analysis; Mean Difference (Net) = 0.02, Standard Error of Mean 0.09

127. Secondary Outcome: Self-efficacy to Use a Dental Dam
Description: as for outcome 125
Time Frame: 12 month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Media Aware for Young Adults | Delayed Intervention Control | Active Comparator: Active Control - Health Aware for Young Adults
Number analyzed (Participants) | 551 | 588 | 508
score on a scale | 2.45 (0.06) | 2.37 (0.05) | 2.32 (0.06)
Statistical Analysis 1: Comparison: Intervention - Media Aware for Young Adults vs Delayed Intervention Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.277, Mixed Models Analysis; Mean Difference (Net) = 0.08, Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Intervention - Media Aware for Young Adults vs Active Comparator: Active Control - Health Aware for Young Adults; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.115, Mixed Models Analysis; Mean Difference (Net) = 0.14, Standard Error of Mean 0.09

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from pretest to last follow-up completion: approximately 12 months
Arm/Group | Intervention - Media Aware for Young Adults | Active Control - Health Aware for Young Adults | Delayed Intervention Control
All-Cause Mortality (participants affected / at risk) | 0/551 | 0/508 | 0/588
Serious Adverse Events (participants affected / at risk) | 0/551 | 0/508 | 0/588
Other Adverse Events (participants affected / at risk) | 0/551 | 0/508 | 0/588

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT04950686/Prot_SAP_000.pdf